CLINICAL TRIAL: NCT06490601
Title: Long Term Comparison of Combination Therapy (Thalidomide and Hydroxyurea) vs Thalidomide Alone in Beta Thalassemia.
Brief Title: Long Term Beta Thalassemia Treatment: Findings From The Extension Period
Acronym: Thalidomide
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Blood and Marrow Transplant (NIBMT), Pakistan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIBD/IRB-242/12-2022
Record Dates: First submitted 2024-06-21; First posted 2024-07-08 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Fetal Hemoglobin; Beta-Thalassemia; Hemoglobinopathies
Keywords: thalidomide; safety and efficacy; thalassemia; fetal hemoglobin inducer; hydroxyurea
MeSH Terms: conditions — beta-Thalassemia; Hemoglobinopathies; Thalassemia | interventions — Thalidomide; Hydroxyurea; Combined Modality Therapy

STUDY DESIGN:
Intervention Model Description: study participants were divided into 2 groups. one was treated with combination therapy that includes thalidomide and hydroxyurea whereas another group was treated with thalidomide alone.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- combination therapy (thalidomide and hydroxyurea) (Experimental): In this group, participants were treated with combination therapy that includes thalidomide and hydroxyurea at the dose of 100mg/day at night with aspirin and 500mg /day respectively.
  Interventions: Drug: thalidomide and hydroxyurea
- thalidomide alone (Active Comparator): In this group, participants were treated with thalidomide at the dose of 100mg/day at night with aspirin.
  Interventions: Drug: Thalidomide

INTERVENTIONS:
Drug: thalidomide and hydroxyurea — Thalidomide:
  Thalidomide glutarimide is derivation of glutamic acid. Potentiating of fetal hemoglobin expression occurs by up regulation of Erythroid transcription factor and Erythroid Krüppel-like factor expression Furthermore few studies also concluded that thalidomide hypomethylate 27th amino acid in Histone H3 in the gamma globin gene. Initiating cause of this process is suppression of Nuclear factor (kappa-light-chain-enhancer of activated B cells) activation by tumor necrosis factor- alpha Vascular endothelial growth factor , Prostaglandin E2 and inflammatory cytokine.
  Hydroxyurea:
  Hydroxyurea or hydroxycarbamide (HU) lies in the category of antimetabolite. Mechanism of fetal hemoglobin induction includes increase in erythropoietin and nitric oxide production, apoptosis induction and potentiating in granulocyte cycling activity.
  Other Names: combination therapy in beta thalassemia
  Arms: combination therapy (thalidomide and hydroxyurea)
Drug: Thalidomide — Thalidomide glutarimide is derivation of glutamic acid. Potentiating of fetal hemoglobin expression occurs by up regulation of Erythroid transcription factor and Erythroid Krüppel-like factor expression Furthermore few studies also concluded that thalidomide hypomethylate 27th amino acid in Histone H3 in the gamma globin gene. Initiating cause of this process is suppression of Nuclear factor (kappa-light-chain-enhancer of activated B cells) activation by tumor necrosis factor -alpha , Vascular endothelial growth factor , Prostaglandin E2 and inflammatory cytokine.
  Investigating the impact of thalidomide on transfusion-dependent beta thalassemia patients is essential for discerning its therapeutic efficacy and safety profile.
  Other Names: fetal hemoglobin inducer
  Arms: thalidomide alone

SUMMARY:
The project, titled "Long Term Beta Thalassemia Treatment: Findings From The Extension Period Of Phase 2 Clinical Trial," aims to compare the efficacy and safety of combination therapy (thalidomide and hydroxyurea) versus thalidomide alone. The study, lasting three years, is a Phase 2 single-center, open-label interventional study with a sample size of 30 participants aged 8-35 years. It includes specific inclusion and exclusion criteria for participant selection. Data will be collected through clinical interviews and medical records and analyzed using(Statistical Package for the Social Sciences. This project aims to enhance beta thalassemia treatment strategies, focusing on reducing transfusion dependency and improving patient quality of life.

DETAILED DESCRIPTION:
Study titled Long Term Beta Thalassemia Treatment: Findings From The Extension Period Of Phase 2 Clinical Trial, conducted at the National Institute of Blood Disease & Bone Marrow Transplantation (NIBD & BMT).

This study focuses on the long-term comparison of combination therapy (thalidomide and hydroxyurea) versus thalidomide alone in treating beta thalassemia. The objective is to evaluate the efficacy and safety of the combination therapy compared to thalidomide alone, with the hypothesis that the combination will be more effective. Beta thalassemia is defined as an autosomal recessive disorder affecting beta-globin production, influenced by genetic modifiers. Key variables include hemoglobin, red blood cells, leukocyte count, reticulocyte count, platelets, lactate dehydrogenase, nucleated red blood cells, ferritin, bilirubin, Serum Glutamate Pyruvate Transaminase, creatinine, transfusion frequency, spleen and liver size, hemoglobin subunit beta [ Homo sapiens (human) ] mutation, and certain polymorphism in gamma globin gene . The study took place at NIBD hospital over three years, designed as a Phase 2 single-center, two-arm open-label interventional study with a sample size of 30 participants using simple randomized sampling. Inclusion criteria are beta thalassemia major/intermediate patients aged 8-35 years, while exclusion criteria include patients with liver dysfunction, married patients, lactating mothers, and those with a history of thrombosis and fits. Data will be collected through clinical interviews and medical record reviews and analyzed using (Statistical Package for the Social Sciences.

ELIGIBILITY:
Inclusion Criteria:

* Known case of beta thalassemia major/intermediate (transfusion dependent)
* Willing to give informed consent

Exclusion Criteria

* Patients with comorbidities such as liver dysfunction
* Married patients
* Lactating mothers
* History of thrombosis and fits

Ages: 8 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
hemoglobin levels | 3 years
  Measure the improvement in hemoglobin levels Hemoglobin levels will be assessed using a complete blood count (CBC) test, measured in grams per deciliter (g/dL) of blood. This test is conducted through a venous blood sample, which is then analyzed using an automated hematology analyzer to determine the hemoglobin concentration.
red blood cell count. | 3 years
  Measure the improvement in red blood cell count. Red blood cell count will be assessed using a complete blood count (CBC) test, measured in millions of cells per microliter (million cells/µL) of blood. This test is conducted through a venous blood sample, analyzed using an automated hematology analyzer to determine the number of red blood cells present.
leukocyte count | 3 years
  Measure the effect on in leukocyte count Leukocyte count will be assessed using a complete blood count (CBC) test, measured in thousands of cells per microliter (thousand cells/µL) of blood. This test involves analyzing a venous blood sample with an automated hematology analyzer to determine the total number of white blood cells present.
reticulocyte count | 3 years
  Measure the effect on reticulocyte count Reticulocyte count will be assessed using a complete blood count (CBC) test, measured as a percentage of the total red blood cells or as an absolute number per microliter (µL) of blood. This test involves analyzing a venous blood sample with an automated hematology analyzer, which identifies and quantifies reticulocytes using specific staining techniques.
Transfusion Frequency: | 3 years
  Document and compare the frequency of blood transfusions required by patients in both treatment arms over the study period.
  Transfusion frequency will be assessed by recording the number of blood transfusions a patient receives over a specified period, such as weekly, monthly, or annually. This data will be collected from patient medical records and/or transfusion logs, ensuring accurate tracking of each transfusion event.

SECONDARY OUTCOMES:
Spleen and Liver Size | 3 years
  Measure changes in spleen and liver size as a response to the treatments. Spleen and liver size will be assessed using imaging techniques such as ultrasound.. Measurements will be reported in centimeters (cm), capturing the dimensions of each organ to evaluate any enlargement or abnormalities.
Serum Ferritin Levels | 3 years
  Evaluate the effectiveness of the combination therapy in reducing serum ferritin levels, indicating decreased iron overload.
  Serum ferritin levels will be assessed using a blood test, measured in nanograms per milliliter (ng/mL). A venous blood sample will be analyzed in a clinical laboratory using immunoassay techniques to determine the concentration of ferritin, providing an indicator of the body's iron stores.
Genetic Modifiers: | 3 years
  Analyze the influence of genetic modifiers. Genetic modifiers will be assessed through genetic testing,e.g thalassemia genetic profile focusing on specific genes or genetic variations known to influence the expression or function of proteins related to the condition under study. This analysis helps identify how genetic factors may modify disease progression, treatment response, or other relevant outcomes.
bilirubin | 3 years
  Monitor and compare changes in biochemical parameters such as bilirubin. Bilirubin levels will be assessed through a blood test, typically measured in milligrams per deciliter (mg/dL). This test analyzes a venous blood sample to determine the concentration of bilirubin, a pigment produced from the breakdown of red blood cells, providing insights into liver function and potential health conditions such as jaundice or liver disease.
lactate dehydrogenase. | 3 years
  Monitor and compare changes in biochemical parameters such as lactate dehydrogenase.
  Lactate dehydrogenase (LDH) levels will be assessed through a blood test, measured in units per liter (U/L). This test analyzes a venous blood sample to determine the concentration of LDH, an enzyme involved in cellular metabolism. Elevated LDH levels may indicate tissue damage or disease.
Serum Glutamate Pyruvate Transaminase, | 3 years
  Monitor and compare changes in biochemical parameters such as Serum Glutamate Pyruvate Transaminase. Serum Glutamate Pyruvate Transaminase, also known as alanine aminotransferase (ALT), will be assessed through a blood test, measured in units per liter (U/L). This test analyzes a venous blood sample to determine the concentration of ALT, an enzyme primarily found in the liver cells. Elevated ALT levels may indicate liver damage or disease.
creatinine | 3 years
  Monitor and compare changes in biochemical parameters such as creatinine. Creatinine levels will be assessed through a blood test, typically measured in milligrams per deciliter (mg/dL) or micromoles per liter (µmol/L). This test involves analyzing a venous blood sample to determine the concentration of creatinine, a waste product from muscle metabolism filtered by the kidneys. Monitoring creatinine levels helps evaluate kidney function and detect conditions such as kidney disease or impaired renal function.

OTHER OUTCOMES:
Safety Profile: | 3 years
  Assess the safety and tolerability of the combination therapy versus thalidomide alone by monitoring adverse effects and clinical complications.
  The safety profile will be assessed by monitoring and documenting adverse events, side effects, and any other safety-related outcomes throughout the study period. This includes recording and analyzing data on patient-reported symptoms, clinical observations, laboratory test results (including those for the parameters previously discussed like liver enzymes, kidney function tests, etc.), and any other relevant safety assessments specified in the study protocol.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of blood disease and bone marrow transplant, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
it will decide later.

REFERENCES:
- [Background] Henson DE. Loss of p53-immunostaining intensity in breast cancer. J Natl Cancer Inst. 1996 Aug 7;88(15):1015-6. doi: 10.1093/jnci/88.15.1015. No abstract available. PMID 8683628